CLINICAL TRIAL: NCT03347604
Title: Effect of Body Position on Spirometry in Abdominal Obesity.
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Antranik Mangardich, Medical Doctor, Rush University Medical Center
Other Study IDs: ORA: 17060206-IRB01
Record Dates: First submitted 2017-10-24; First posted 2017-11-20 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with abdominal obesity: Enrolling patients with abdominal obesity as defined by WHO to have waist to hop ratio of > 0.85 in women, or > 0.9 in men.
  Interventions: Diagnostic Test: Supine spirometry, MIPs and MEPs

INTERVENTIONS:
Diagnostic Test: Supine spirometry, MIPs and MEPs — We are going to test spirometry while in supine position , and also test respiratory muscles by measuring the maximum inspiratory and maximum expiratory efforts made by patients.

SUMMARY:
Objective: Study the effect of body position on spirometry in obese patients as defined by waist to hip ratio (WHR) of greater than 0.85 in women, and 0.9 in men

Background: Spirometry is routinely ordered to work up dyspnea in obesity. The most common abnormality is a restrictive disease pattern. The underlying mechanisms of this pattern are not completely understood. One plausible explanation is diaphragmatic weakness or skeletal muscle weakness. The change in forced vital capacity (FVC) from sitting to supine is a very sensitive and specific test for detecting diaphragmatic weakness. The effect of body position on spirometry in obesity has not been extensively studied, and there are no studies that look at this when obesity is measured by waist to hip ratio. Effect of body position has been studied in normal patients, and it is expected the FVC can decrease as much as 10% when changing from sitting to supine. The investigators do not know what would be considered 'the normal' amount for FVC to decrease by in the obese population, and thus would like to test patients with increased WHR both in sitting and supine position. The investigators also want to do muscle strength test by measuring the maximal inspiratory and expiratory pressures (MIPs and MEPs).

Anticipated results: the investigators anticipate that our study population will replicate the restrictive disease pattern usually seen in obesity. The investigators also anticipate for the FVC to decrease when in the supine position compared to sitting. The amount by which it decreases will likely fall between 10 -25%. The investigators anticipate to not find any abnormalities in MIPs and MEPs in obesity.

DETAILED DESCRIPTION:
The design for this study will be a cross-sectional study. This study will be conducted in the pulmonary function laboratory at Rush University Medical Center. A sample of subjects who meet the inclusion criteria will be selected from the adult population scheduled for CPFT lab appointments. The details of the study will be discussed by the respiratory therapist prior to the end of CPFT study. Information normally gathered in routine CPFTs includes oxygen saturation, height, and weight. Additional measures for subjects who accept the invitation to participate in this study will include measurements of BMI, waist circumference, and hip circumference. Inclusion criteria includes individuals of both genders, age of 18 years or older and individuals with abdominal obesity as defined by WHO as WHR greater than 0.85 in women, and 0.90 in men. Exclusion criteria include patients who cannot understand or comply with the spirometry test, known lung disease, obstructive ventilatory defect on CPFT, chest wall abnormalities/disorders, known neuromuscular disease, pregnant patients or prisoners.

The BMI (kg/m2) will be calculated as weight (in kilograms) divided by square of the height (in meters). Waist-hip ratio (WHR) will be measured in the standing position using a stretch-resistant tape. Waist circumference will be measured at a midpoint between the lowest rib and the middle of the iliac crest. The hip is defined as the maximal circumference around the gluteal muscles below the iliac crests.8,9 These measurements will be obtained by respiratory therapists who have been trained in obtaining WHR measurements using a standardized patient to assure measurement fidelity.

Spirometry measurements of FEV1 and FVC will be made in two testing positions for this study; the patients seated 90o upright (sitting position), and the patient fully supine position (0º horizontal decubitus position). FVC (forced vital capacity) is the volume of air in liters that can be forcibly and maximally exhaled after taking in the deepest breath. FEV1 is the volume of air that can be forcibly exhaled from the lungs in the first second of a forced expiratory maneuver and is reported in liters. Lung volumes will also be measured in the sitting position using either body plethysmography or nitrogen washout method as part of the routine CPFT testing. Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), will also be measured in the sitting position and reported in centimeters of water (cm H2O). These reflect the maximum pressures generated by the patient on inhalation and exhalation, respectively and test respiratory muscle strength. All tests will be conducted in accordance with 2005 American Thoracic Society/European Respiratory Society guidelines13 using the Sensormedics Vmax pulmonary function system. The Vmax system is calibrated daily and reports all measurements at body temperature, pressure and water vapor. All tests will be performed by a team of respiratory therapists who have demonstrated annual competence following the recommendations of the American Thoracic Society/European Respiratory Society.14

Individuals who meet the study criteria and are able to successfully complete a CPFT will be recruited to participate in the study. After completing a consent form, the waist and hip measurements will be made. MIP and MEP measures will be made in the sitting position. Testing of spirometry will be repeated in the supine position. Sitting FEV1, FEV1 % predicted, FVC, FVC % predicted, FEV1/SVC, lower limit of normal for FEV1/FVC, supine FEV1, FEV1 % predicted, FVC, FVC % predicted, MIP, MEP, ERV, RV, FRC and TLC will be extracted from the pulmonary function test results and entered in REDCap for data tracking. Age, race, gender, and diagnosis code will be taken from the information routinely gathered for a pulmonary function test. The question related to smoking history will be asked directly of the subject. All data will be entered into REDCap.

Procedures done for research purposes and procedures done for routine clinical management:

A routine complete pulmonary function test (CPFT) as ordered by their referring provider includes measurements of slow vital capacity by spirometry, forced vital capacity by spirometry, lung diffusion by DLCO, and measurement of lung volume by body plethysmography. All of these measurements will be performed while the patient in sitting position. The additional testing for this study includes spirometry while the patient is in the supine position; and MIPs, and MEPs in the sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders, age of 18 years or older
* Individuals with abdominal obesity with WHR > 0.85 in women, > 0.9 in men
* Ability of patients to transfer themselves into a cardiac chair
* Able to understand and comply with testing instructions

Exclusion Criteria:

* Patients who are less than 18 years old
* Patients who are unable to perform an acceptable and repeatable forced vital capacity
* Airflow limitation as evidenced by sitting FEV1/VC < lower limit of normal
* Patients who have a WHR < 0.85 in women, or < 0.9 in men
* Patients who become lightheaded during sitting spirometry
* Patients who cannot transfer themselves independently to a cardiac chair
* History of lung disease (known obstructive or restrictive lung disease)
* Chest wall abnormalities or kyphoscoliosis
* Neuromuscular disease
* Active hemoptysis or recent angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is 30 medically stable obese patients with WHR > 0.85 in women, or > 0.9 in men, coming to outpatient clinic at Rush University Medical Center for complete pulmonary function testing.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1, unit is Liters) | first and only visit in study
  Investigators will measure FEV1 for patient in ight position.
Forced vital capacity (FVC , unit is Liters) | first and only visit in study
  Investigators with measure FVC in upright position.
Forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) | first and only visit in study
  Ratio of FEV1/FVC in supine position.
Total lung capacity (TLC, unit is Liters). | first and only visit in study
  Investigators will measure TLC in upright position.
Maximum inspiratory pressure (MIP, unit is cm of water). | first and only visit in study
  Investigators will measure MIP in upright position.
Maximum expiratory pressure (MEP, unit is cm of water). | first and only visit in study
  Investigators will measure MEP in upright position.
Forced vital capacity (FVC , unit is L) | first and only visit in study
  Does supine position decrease forced vital capacity in abdominal obese ? Investigators will measure FVC in supine/lying down position.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuczmarski RJ, Flegal KM, Campbell SM, Johnson CL. Increasing prevalence of overweight among US adults. The National Health and Nutrition Examination Surveys, 1960 to 1991. JAMA. 1994 Jul 20;272(3):205-11. doi: 10.1001/jama.272.3.205. PMID 8022039
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Guilbert JJ. The world health report 2002 - reducing risks, promoting healthy life. Educ Health (Abingdon). 2003 Jul;16(2):230. doi: 10.1080/1357628031000116808. No abstract available. PMID 14741909
- [Background] Wing RR, Matthews KA, Kuller LH, Meilahn EN, Plantinga P. Waist to hip ratio in middle-aged women. Associations with behavioral and psychosocial factors and with changes in cardiovascular risk factors. Arterioscler Thromb. 1991 Sep-Oct;11(5):1250-7. doi: 10.1161/01.atv.11.5.1250. PMID 1911710
- [Background] Saxena Y, Sidhwani G, Upmanyu R. Abdominal obesity and pulmonary functions in young Indian adults: a prospective study. Indian J Physiol Pharmacol. 2009 Oct-Dec;53(4):318-26. PMID 20509323
- [Background] Harik-Khan RI, Wise RA, Fleg JL. The effect of gender on the relationship between body fat distribution and lung function. J Clin Epidemiol. 2001 Apr;54(4):399-406. doi: 10.1016/s0895-4356(00)00318-8. PMID 11297889
- [Background] Al Ghobain M. The effect of obesity on spirometry tests among healthy non-smoking adults. BMC Pulm Med. 2012 Mar 21;12:10. doi: 10.1186/1471-2466-12-10. PMID 22436173
- [Background] Koenig SM. Pulmonary complications of obesity. Am J Med Sci. 2001 Apr;321(4):249-79. doi: 10.1097/00000441-200104000-00006. PMID 11307867
- [Background] TUCKER DH, SIEKER HO. The effect of change in body position on lung volumes and intrapulmonary gas mixing in patients with obesity, heart failure, and emphysema. Am Rev Respir Dis. 1960 Dec;82:787-91. doi: 10.1164/arrd.1960.82.6.787. No abstract available. PMID 13778537
- [Background] BLAIR E, HICKAM JB. The effect of change in body position on lung volume and intrapulmonary gas mixing in normal subjects. J Clin Invest. 1955 Mar;34(3):383-9. doi: 10.1172/JCI103086. No abstract available. PMID 14354008
- [Background] Shimokata H, Andres R, Coon PJ, Elahi D, Muller DC, Tobin JD. Studies in the distribution of body fat. II. Longitudinal effects of change in weight. Int J Obes. 1989;13(4):455-64. PMID 2676875
- [Background] Sievenpiper JL, Jenkins DJ, Josse RG, Leiter LA, Vuksan V. Simple skinfold-thickness measurements complement conventional anthropometric assessments in predicting glucose tolerance. Am J Clin Nutr. 2001 Mar;73(3):567-73. doi: 10.1093/ajcn/73.3.567. PMID 11237933
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Lung function testing: selection of reference values and interpretative strategies. American Thoracic Society. Am Rev Respir Dis. 1991 Nov;144(5):1202-18. doi: 10.1164/ajrccm/144.5.1202. No abstract available. PMID 1952453
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Ceylan E, Comlekci A, Akkoclu A, Ceylan C, Itil O, Ergor G, Yesil S. The effects of body fat distribution on pulmonary function tests in the overweight and obese. South Med J. 2009 Jan;102(1):30-5. doi: 10.1097/SMJ.0b013e31818c9585. PMID 19077765
- [Background] Chen Y, Rennie D, Cormier YF, Dosman J. Waist circumference is associated with pulmonary function in normal-weight, overweight, and obese subjects. Am J Clin Nutr. 2007 Jan;85(1):35-9. doi: 10.1093/ajcn/85.1.35. PMID 17209174
- [Background] Domingos-Benicio NC, Gastaldi AC, Perecin JC, Avena KM, Guimaraes RC, Sologuren MJ, Lopes-Filho JD. [Spirometric values of obese and non-obese subjects on orthostatic, sitting and supine positions]. Rev Assoc Med Bras (1992). 2004 Apr-Jun;50(2):142-7. doi: 10.1590/s0104-42302004000200028. Epub 2004 Jul 21. Portuguese. PMID 15286860
- [Background] Magnani KL, Cataneo AJ. Respiratory muscle strength in obese individuals and influence of upper-body fat distribution. Sao Paulo Med J. 2007 Jul 5;125(4):215-9. doi: 10.1590/s1516-31802007000400004. PMID 17992391
- [Background] Al-Bader WR, Ramadan J, Nasr-Eldin A, Barac-Nieto M. Pulmonary ventilatory functions and obesity in Kuwait. Med Princ Pract. 2008;17(1):20-6. doi: 10.1159/000109585. PMID 18059096
- [Background] Bae J, Ting EY, Giuffrida JG. The effect of changes in the body position obsese patients on pulmonary volume and ventilatory function. Bull N Y Acad Med. 1976 Sep;52(7):830-7. No abstract available. PMID 1066179
- [Background] Vilke GM, Chan TC, Neuman T, Clausen JL. Spirometry in normal subjects in sitting, prone, and supine positions. Respir Care. 2000 Apr;45(4):407-10. PMID 10780036
- [Background] Lechtzin N, Wiener CM, Shade DM, Clawson L, Diette GB. Spirometry in the supine position improves the detection of diaphragmatic weakness in patients with amyotrophic lateral sclerosis. Chest. 2002 Feb;121(2):436-42. doi: 10.1378/chest.121.2.436. PMID 11834654
- [Background] Fromageot C, Lofaso F, Annane D, Falaize L, Lejaille M, Clair B, Gajdos P, Raphael JC. Supine fall in lung volumes in the assessment of diaphragmatic weakness in neuromuscular disorders. Arch Phys Med Rehabil. 2001 Jan;82(1):123-8. doi: 10.1053/apmr.2001.18053. PMID 11239298
- [Background] Teixeira AB, Mathias LA, Saad Junior R. The influence of posture on spirometric values in grade III obese patients. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):713-9. doi: 10.1016/S0034-7094(11)70080-0. English, Multiple languages. PMID 22063372